CLINICAL TRIAL: NCT02537327
Title: Epidemiological Study on the Incidence and Characteristics of Secondary Caries Next to Tooth Restorations
Brief Title: Incidence of Recurrent Caries Next to Tooth Restorations
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S56046
Record Dates: First submitted 2015-08-19; First posted 2015-09-01 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-06

CONDITIONS: Recurrent Caries
Keywords: Recurrent caries; Secondary caries; Dental composite; Dental amalgam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to determine the incidence of recurrent caries around the different types of restorative materials (composites, amalgam, ceramics, crowns, etc.) and to better characterize recurrent caries lesions in terms of location and size of the lesions and type, material and age of the restoration.

DETAILED DESCRIPTION:
The data will be collected from patients who are visiting the dental clinic for a check-up. These data will be retrieved in the patient records. In particular the clinical (mouth) exam and the radiographic images ('RX-bite-wings'), which are routinely taken during these check-up consultations, will be used for the evaluation of recurrent caries. Information regarding medical background, oral hygiene, sugar eating habits and possible parafunctional activities will also be gathered from the patient files. In addition, caries risk of the patients will be assessed using commercial kits for analysis of their saliva (Saliva-Check Buffer, GC, Tokyo, Japan) and dental plaque (Tri Plaque ID Gel, GC, Tokyo, Japan), which are a part of the routine care of the patients at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting the university dental clinic (Department of Oral Health Care) for a dental check-up

Exclusion Criteria:

* Patients for who not all necessary data could be registered (incomplete mouth exam records, missing RX-bite wings, etc)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting the university dental clinic (Department of Oral Health Care) for a dental check-up
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2014-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of recurrent caries | Two years
  Number of recurrent caries lesions (new caries lesion next to restoration) within a specified time period divided by the total number of restorations.

SECONDARY OUTCOMES:
Caries risk of the patient | Two years
  Caries risk of each patient will be assessed based on scoring of several parameters such as: number of new caries lesions in the last 3 years (from patients' files), presence of relevant systemic disease (from patients' files), sugar consumption (from patients' files), oral hygiene (from patients' files) and results of the Saliva-check test and Tri plaque ID test.

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten L. Van Landuyt, DDS, PhD, Study Chair — BIOMAT, Department of Oral Health Sciences, University of Leuven & Dentistry University Hospitals Leuven
Locations (1):
- KU Leuven and UZ Leuven, Department of oral health sciences, Leuven, Belgium